CLINICAL TRIAL: NCT00795756
Title: A Randomized Study on CNS Prophylaxis With Liposome-Encapsulated Cytarabine in Association With a Lineage-Targeted and MRD-Oriented Postremission Strategy in Adult ALL
Brief Title: Intrathecal DepoCyte and Lineage-targeted Minimal Residual Disease-oriented Therapy of Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northern Italy Leukemia Group (Other)
Responsible Party: Principal Investigator, DR RENATO BASSAN, Medical Doctor, Northern Italy Leukemia Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NILG-ALL 10/07
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Adults; Central nervous system prophylaxis; Minimal residual disease
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — Methotrexate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrathecal DepoCyte (Experimental): I.t. DepoCyte 50 mg admninistered x6-8 (depending on immunophenotypic disease subset) during induction/consolidation/eraly maintenance phases
  Interventions: Drug: liposome-encapsulated cytarabine (DepoCyte)
- Triple intrathecal therapy (TIT) (Active Comparator): Methotrexate 12,5 mg + Cytarabine 50 mg + Prednisolone 40 mg injected intrathecally x12 during indiction/consolidation phases
  Interventions: Drug: Triple intrathecal therapy (TIT)

INTERVENTIONS:
Drug: liposome-encapsulated cytarabine (DepoCyte) — DepoCyte 50 mg injected intrathecally x6-8 (6: B-lineage, 8: T-lineage) during induction/consolidation phases
  Other Names: DepoCyte; DepoCyt
  Arms: Intrathecal DepoCyte
Drug: Triple intrathecal therapy (TIT) — Methotrexate 12,5 mg + Cytarabine 50 mg + Prednisolone 40 mg. injected intrathecally x12 during induction/consolidation therapy
  Other Names: Methotrexate; Cytosine arabinoside; Cytosar
  Arms: Triple intrathecal therapy (TIT)

SUMMARY:
The aim of this clinical study in adult ALL is to compare by risk category (1) the feasibility of two different CNS prophylaxis regimens and (2) the overall disease-free survival in relation to the achievement of an early MRD negative status and following consolidation with lineage-targeted methotrexate infusions and other disease-specific therapeutic elements, with or without the application of allogeneic or autologous SCT depending on risk class and MRD study results.

In this multicentric prospective pilot randomized phase II trial on CNS prophylaxis, all patients receive induction/consolidation therapy incorporating lineage-targeted high-dose methotrexate plus other drugs (with additional imatinib in Ph/BCR-ABL+ ALL), for the achievement of an early negative MRD status. The MRD study supports a risk/MRD-oriented final consolidation phase.

DETAILED DESCRIPTION:
A) Risk Classification

Newly diagnosed patients are hierarchically clustered into very high, high and standard risk cases (VHR, HR, SR) using international risk criteria modified according to NILG:

A1) VHR (any criterium): B-precursor: WBC count >100x109/L; adverse cytogenetics/molecular biology such as t(9;22)/BCR-ABL, t(4;11)/MLL rearrangement at 11q23, +8, -7, del6q, t(8;14), low hypodiploidy with 30-39 chromosomes, near triploidy with 60-78 chromosomes, complex with >5 unrelated anomalies. T-precursor: WBC count >100x109/L; early/late non-cortical immunophenotype (CD1a-); adverse cytogenetics/molecular biology (as above).

A2) HR (any criterium, VHR excluded): B-precursor: WBC count >30x109/L; pro-B immunophenotype; complete remission after cycle 2. T-precursor: complete remission after cycle 2.

A3) SR (all criteria, VHR/HR excluded): B-precursor: WBC count <30x109/L; T-precursor: WBC count <100x109/L; cortical immunophenotype (CD1a+).

B) CNS Prophylaxis Stratification before randomisation

1. by immunophenotype, i.e. B-precursor vs. T-precursor
2. by risk class, i.e. SR vs. non-SR (using only known factors) Randomisation: intrathecal (IT) CNS prophylaxis with standard triple therapy (TIT, 12 total injections) vs. DepoCyte (6-8 total injections by disease subset). Cranial irradiation is omitted in both arms, and all patients receive the same chemotherapy program including CNS-crossing agents.

C)Induction/Early Consolidation and MRD Study

Randomised patients receive homogeneous induction/early consolidation chemotherapy, including subset-specific elements for B-precursor ALL (3x targeted-infusion methotrexate 2.5 g/m2), T-precursor ALL (3x targeted-infusion methotrexate 5 g/m2), age >55 years (methotrexate reduced to 1.5 g/m2), Ph/BCR-ABL+ ALL (imatinib, reduced-intensity chemotherapy), radiation therapy (LL). Patients not in CR after cycles 1-2 are off study. For CR evaluation bone marrow is checked on days 28 and/or 56. Consolidation cycles are administered at 21-28 day intervals Concurrent MRD analysis is performed at four timepoints (weeks 4, 10, 16 and 22 of induction/consolidation), to optimize risk classification and support risk/MRD-oriented therapy:

C1) MRD negative (M-NEG): negative MRD study (<10-4 at timepoints #2 and #3, and negative at timepoint #4) C2) MRD positive (M-POS): positive MRD study (>10-4 at timepoints #2 or #3, or positive at timepoint #4)

D)MRD/Risk-Oriented Final Therapy D1) VHR patients are candidate to an early allogeneic SCT (related/unrelated donor/cord blood; ablative/non-ablative conditioning according to current protocols/guidelines) after CR, regardless MRD study results.

D2) M-POS as well as HR patients with unknown MRD are allocated to allogeneic SCT after MRD timepoint 2 (M-POS >10-4) or MRD timepoint 4 (others). When an allogeneic SCT is not possible, patients complete consolidation and receive autologous-type SCT followed by maintenance.

D3) M-NEG as well as SR patients with unknown MRD are allocated to maintenance therapy.

Age-limited therapeutic procedures: Patients aged >55 years are treated with age-adapted therapy, and when indicated will be included in SCT programs whenever possible and according to performance status and comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Diagnosis of untreated ALL with B-/T-precursor phenotype or B-cell lymphoblastic lymphoma (B-LL), either de novo or secondary to chemo-radiotherapy for other cancer.
* Full cytological, cytochemical, cytogenetic and immunobiological disease characterization by revised FAB, EGIL and WHO criteria.
* Bone marrow and peripheral blood sampling (ALL) or biopsy specimen (LL) for MRD study.
* ECOG performance status 0-2 or reversible ECOG 3 score following intensive care of complications.
* Signed informed consent.

Exclusion Criteria:

* Diagnosis of B-ALL (FAB L3 ALL/Burkitt's leukemia or lymphoma) and T-LL (T-cell lymphoblastic lymphoma).
* Down's syndrome.
* Pre-existing, uncontrolled pathology such as cardiac disease (congestive/ischemic, acute myocardial infarction within the past 3 months, untreatable arrythmias, NYHA classes III and IV), severe liver disease with serum bilirubin >3 mg/dL and/or ALT >3 x upper normal limit (unless attributable to ALL/LL), kidney function impairment with serum creatinine >2 mg/dL (unless attributable to ALL/LL), and severe neurological or psychiatric disorder that impairs the patient's ability to understand and sign the informed consent, or to cope with the intended treatment plan.
* Known HIV positive serology.
* Other active hematological or non-hematological cancer with life expectancy <1 year.
* Pregnancy (fertile women will be advised not to become pregnant while on treatment; and male patients to adopt contraceptive methods), unless therapeutic aborption/early discharge is carried out.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2008-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Comparative analysis of feasibility/toxicity of IT DepoCyte vs. TIT | weeks 5, 11, 17 and 23

SECONDARY OUTCOMES:
Comparative analysis of isolated and combined CNS recurrence following TIT vs DepoCyte prophylaxis | During study follow-up
Complete remission (CR) | After study chemotherapy cycles 1 and 2
Bone marrow MRD negativity rates | Four time-points at weeks 4-22
Lenght of remission | Study follow-up
Overall survival | Study follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Renato Bassan, MD, Study Chair — USC Ematologia, Ospedali Riuniti, Bergamo (Italy)
Locations (16):
- Italy (16):
  - USC Ematologia, Ospedale Civile, Alessandria, (al)
  - USC Ematologia, Ospedali Riuniti, Bergamo, (bg)
  - Divisione di Ematologia - Spedali Civili, Brescia, (bs)
  - Divisione di Ematologia e TMO, Ospedale San Maurizio, Bolzano, (bz)
  - Ematologia e centro TMO - Ospedale Armando Businco, Cagliari, (ca)
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo, (cn)
  - Ematologia e centro TMO, Istituti Ospedalieri, Cremona, (cr)
  - Ematologia - AOU Careggi, Florence, (fi)
  - Ematologia e centro TMO - IRCSS Mangiagalli Regina Elena, Milan, (mi)
  - Ematologia e centro TMO, Ospedale San Raffaele, Milan, (mi)
  - Ematologia e centro TMO, Ospedale San Gerardo, Monza, (mi)
  - Oncoematologia e TMO - Dipartimento Oncologico La Maddalena, Palermo, (pa)
  - Ematologia 2 - Ospedale San Giovanni Battista, Torino, (to)
  - Medicina Interna I - Ospedale di Circolo, Varese, (va)
  - Onco-Ematologia - Ospedale Civile, Noale, (ve)
  - Ematologia - Ospedale San Bortolo, Vicenza, (vi)

REFERENCES:
- [Derived] Bassan R, Masciulli A, Intermesoli T, Audisio E, Rossi G, Pogliani EM, Cassibba V, Mattei D, Romani C, Cortelezzi A, Corti C, Scattolin AM, Spinelli O, Tosi M, Parolini M, Marmont F, Borlenghi E, Fumagalli M, Cortelazzo S, Gallamini A, Marfisi RM, Oldani E, Rambaldi A. Randomized trial of radiation-free central nervous system prophylaxis comparing intrathecal triple therapy with liposomal cytarabine in acute lymphoblastic leukemia. Haematologica. 2015 Jun;100(6):786-93. doi: 10.3324/haematol.2014.123273. Epub 2015 Mar 6. PMID 25749825